CLINICAL TRIAL: NCT00765635
Title: Randomized, Placebo-Controlled Evaluation of Chlorobutanol, Potassium Carbonate, and Irrigation in Cerumen Removal
Brief Title: Chlorobutanol, Potassium Carbonate, and Irrigation in Cerumen Removal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Miguel Caballero / ENT specialist, Hospital clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLO2008/4503
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-10

CONDITIONS: Ear Infection; Hearing Loss; Vertigo
Keywords: complete occlusion of the ear canal due to cerumen
MeSH Terms: conditions — Otitis; Hearing Loss; Vertigo | interventions — Otocerum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 (Experimental): Taponoto ® (potassium carbonate 20 mg/1 ml, ethyl alcohol, glycerol 480, thymol 0.4; Teofarma Iberica S.A., Barcelona, Spain),
  Interventions: Drug: drops intilation (Taponoto ® )
- 3 (Placebo Comparator): sterile saline solution (NaCl 0.9%, Braun Medical SA, Barcelona, Spain).
  Interventions: Drug: drops intilation (Placebo)
- 1: Chlorobutanol (Experimental): ceruminolytic product, Otocerum® (Chlorobutanol 50 mg/1 ml, phenol 10 mg/1 ml, turpentine essence 0.15 ml/1 ml, ethyl alcohol; Reig Jofre laboratories, Barcelona, Spain),
  Interventions: Drug: drops intilation (Otocerum®)

INTERVENTIONS:
Drug: drops intilation (Taponoto ® ) — four drops, unique doses
  Arms: 2
Drug: drops intilation (Otocerum®) — four drops, unique doses
  Arms: 1: Chlorobutanol
Drug: drops intilation (Placebo) — Placebo
  Arms: 3

SUMMARY:
Accumulation of cerumen in the external ear canal is a common problem. The presence of cerumen not only interferes with the clinician's view of the tympanic membrane, but may also result in hearing loss and vertigo, and may predispose to ear infections.

Removal of cerumen is facilitated by the use of a variety of ceruminolytics, or wax solvents. The current study was designed to evaluate the ceruminolytic effects of a single, brief application of the two most frequently used products in the investigators area, containing chlorobutanol or potassium carbonate with or without irrigation in the primary care setting in a randomized, single-blind trial. To our knowledge, this is the first randomized study comparing ceruminolytics with chlorobutanol versus potassium carbonate.

DETAILED DESCRIPTION:
INTERVENTIONS: Subjects were randomly assigned to one of three different treatments: Otocerum®; Taponoto ®, and a control group with sterile saline solution (NaCl 0.9%, Braun Medical SA, Barcelona, Spain). The test medication was instilled into an occluded ear for 15 minutes. Following this treatment, the subject's ear was irrigated with 50 mL of water. The main outcome was the proportion of tympanic membranes that were completely visualized after cerumenolytic agents or saline, alone or with irrigation if needed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ear cerumen

Exclusion Criteria:

* Infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
proportion of tympanic membranes that were completely visualized after cerumenolytic agents or saline, alone or with irrigation if needed | 2008

SECONDARY OUTCOMES:
adverse effects | 2008

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, barcelona, Spain

REFERENCES:
- [Background] Roland PS, Eaton DA, Gross RD, Wall GM, Conroy PJ, Garadi R, Lafontaine L, Potts S, Hogg G. Randomized, placebo-controlled evaluation of Cerumenex and Murine earwax removal products. Arch Otolaryngol Head Neck Surg. 2004 Oct;130(10):1175-7. doi: 10.1001/archotol.130.10.1175. PMID 15492164